CLINICAL TRIAL: NCT00366899
Title: A Phase 3, Randomized, Active-Controlled, Double-blind Trial Evaluating the Safety,Tolerability, and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Paediatric Vaccinations in Italy
Brief Title: Study Evaluating a 13-valent Pneumococcal Conjugate Vaccine in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6096A1-500
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Results first posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-01

CONDITIONS: Vaccines, Pneumococcal
Keywords: Vaccine; Infants
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- 2 (Active Comparator): 7-valent pneumococcal conjugate vaccine
  Interventions: Biological: 7 valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — Single 0.5 mL dose of 13vPnC given at 3, 5 and 11 months of age.
  Arms: 1
Biological: 7 valent pneumococcal conjugate vaccine — Single 0.5 mL dose of 7vPnC given at 3, 5 and 11 months of age.
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate (13vPnC) vaccine compared to Prevenar (7vPnC), when given concomitantly with routine paediatric vaccinations in Italy.

ELIGIBILITY:
Inclusion criteria:

1. Aged 3 months (75 to 105 days) at time of enrollment.
2. Available for entire study period and whose parent(s)/legal guardian(s) could be reached by telephone.
3. Healthy infant, as determined by medical history, physical examination, and judgment of the investigator.
4. Born at greater than 32 weeks gestational age and greater than 2000 grams. Regardless of gestational age and birth weight, all subjects must have met inclusion criterion number 3.
5. Parent(s)/legal guardian(s) had to be able to complete all relevant study procedures during study participation.

Exclusion criteria:

1. Previous vaccination with licensed or investigational pneumococcal vaccine.
2. Previous vaccination with Hib conjugate, diphtheria, tetanus, pertussis, polio, or hepatitis B vaccines.
3. A previous anaphylactic reaction to any vaccine or vaccine-related component.
4. Contraindication to vaccination with Hib conjugate, diphtheria, tetanus, pertussis, polio, or hepatitis B, or pneumococcal vaccines.
5. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
6. Known or suspected immune deficiency or suppression.
7. History of culture-proven invasive disease caused by S pneumoniae or Hib.
8. Major known congenital malformation or serious chronic disorder.
9. Significant neurological disorder or history of seizure, including febrile seizure, or significant stable or evolving disorders, such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorders. Did not include resolving syndromes due to birth trauma such as Erb palsy.
10. Receipt of blood products or gamma-globulin (including hepatitis B immunoglobulin and monoclonal antibodies; eg, Synagis® [MedImmune]).
11. Participation in another investigational trial. Participation in purely observational studies was acceptable.
12. Infant who was a direct descendant (eg, child or grandchild) of the study site personnel.

Ages: 75 Days to 105 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 605 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com
Locations (11):
- Italy (11):
  - Taranto, Apulia
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Milan, Lombardy
  - Novara, Piedmont
  - Sassari, Sardinia
  - Palermo, Sicily
  - Ragusa, Sicily
  - Florence, Tuscany

REFERENCES:
- [Derived] Rodgers GL, Esposito S, Principi N, Gutierrez-Brito M, Diez-Domingo J, Pollard AJ, Snape MD, Martinon-Torres F, Gruber WC, Patterson S, Thompson A, Gurtman A, Paradiso P, Scott DA. Immune response to 13-valent pneumococcal conjugate vaccine with a reduced dosing schedule. Vaccine. 2013 Oct 1;31(42):4765-74. doi: 10.1016/j.vaccine.2013.08.009. Epub 2013 Aug 16. PMID 23965217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Italy from October 2006 to March 2007.
Pre-assignment Details: Participants were enrolled into the study according to inclusion/exclusion criteria without a screening period. One subject was prerandomized and counted twice.
Groups:
- 13vPnC: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with diphtheria-tetanus-acellular pertussis (DTPa), hepatitis B, inactivated poliovirus, and hemophilus influenza type b (Hib) vaccine (Infanrix hexa) at 3 and 5 months (infant series), and 11 months of age (toddler dose).
- 7vPnC: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with diphtheria-tetanus-acellular pertussis (DTPa), hepatitis B, inactivated poliovirus, and hemophilus influenza type b (Hib) vaccine (Infanrix hexa) at 3 and 5 months (infant series), and 11 months of age (toddler dose).
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 303 (1 participant was counted twice, 1 participant randomized to 13vPnC, incorrectly received 7vPnC) | 303 (1 participant randomized to 7vPnC but never vaccinated)
Vaccinated Dose 1 | 302 (2 participants randomized to 13vPnC, incorrectly received 7vPnC) | 302
Vaccinated Dose 2 | 296 (1 participant randomized to 13vPnC, incorrectly received 7vPnC) | 293
Completed | 294 | 291
Not Completed | 9 | 12
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Protocol Violation | 2 | 1
Not completed — Failed to return | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Randomized but not consented | 1 | 0
Period: After Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 294 | 291
Completed | 287 | 282
Not Completed | 7 | 9
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 1 | 0
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 287 | 282
Completed | 285 | 281
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 303 | 303 | 606
Age Continuous [Mean (Standard Deviation); unit: months] | 2.9 (0.3) | 2.9 (0.3) | 2.9 (0.3)
Gender [Number; unit: participants] — 1 gender unknown
  participants
    Female | 138 | 133 | 271
    Male | 164 | 170 | 334

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions
Description: Local reactions were collected using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (>7.0 cm). Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: Percentage of Participants
Groups:
- 13vPnC Dose 1: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 3 months of age.
- 7vPnC Dose 1: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 3 months of age.
- 13vPnC Dose 2: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 5 months of age.
- 7vPnC Dose 2: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 5 months of age.
- 13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 11 months of age.
- 7vPnC Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 11 months of age.
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 302 | 302 | 296 | 293 | 294 | 291
Percentage of Participants
  Tenderness - Any (n=234,243,214,215,199,188) | 32.1 | 30.0 | 30.4 | 36.7 | 47.2 | 44.1
  Tenderness-Significant (n=224,231,199,199,164,153) | 2.7 | 3.5 | 4.5 | 5.0 | 8.5 | 5.9
  Swelling - Any (n=232,240,207,209,175,165) | 19.0 | 19.6 | 24.6 | 28.7 | 28.6 | 27.3
  Swelling - Mild (n=232,240,207,208,174,161) | 17.7 | 18.3 | 21.7 | 26.4 | 26.4 | 21.7
  Swelling - Moderate (n=223,229,198,195,160,157) | 3.6 | 3.1 | 5.6 | 5.1 | 7.5 | 10.2
  Swelling - Severe (n=222,229,197,194,159,152) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Redness - Any (n=233,245,213,212,178,174) | 25.8 | 26.5 | 31.5 | 34.4 | 36.5 | 36.2
  Redness - Mild (n=233,244,211,211,178,172) | 24.0 | 24.6 | 28.4 | 32.2 | 32.6 | 30.8
  Redness - Moderate (n=222,231,200,195,160,156) | 2.7 | 3.0 | 5.5 | 3.6 | 7.5 | 10.9
  Redness - Severe (n=243,255,197,194,159,152) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

2. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events
Description: Systemic events (fever ≥ 37.5 degrees Celsius [C], fever ≥ 38 C but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C, decreased appetite, irritability, increased sleep, decreased sleep, hives, use of medication (meds) to treat symptoms, and use of medication to prevent symptoms) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all subjects who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: Percentage of Participants
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 302 | 302 | 296 | 293 | 294 | 291
Percentage of Participants
  Fever ≥38°C but ≤39°C (n=247,246,227,226,204,197) | 41.7 | 38.6 | 55.5 | 60.6 | 63.7 | 52.3
  Fever >39°C but ≤40°C (n=224,233,204,201,167,160) | 3.6 | 4.7 | 6.9 | 7.0 | 9.6 | 12.5
  Fever >40°C (n=222,230,198,195,160,152) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.7
  Decreased appetite (n=246,248,220,218,198,197) | 35.4 | 34.3 | 47.3 | 45.4 | 52.0 | 57.4
  Irritability (n=258,259,245,243,221,227) | 72.9 | 63.7 | 75.5 | 75.3 | 74.7 | 74.9
  Increased sleep (n=269,276,226,232,195,196) | 65.8 | 64.5 | 57.1 | 56.5 | 53.8 | 54.6
  Decreased sleep (n=244,242,222,213,180,171) | 39.3 | 36.4 | 40.1 | 41.8 | 35.6 | 35.7
  Meds-treat symptoms (n=244,245,219,109,192,190) | 34.8 | 30.6 | 43.4 | 47.8 | 53.1 | 43.7
  Meds-prevent symptoms (n=230,238,208,208,172,169) | 12.6 | 18.1 | 20.2 | 24.5 | 27.9 | 24.3

3. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Concomitant Antigen Pertussis, Hepatitis B, Haemophilus Influenzae Type b, Diphtheria, Tetanus and Polio After the 2-Dose Infant Series and After the Toddler Dose
Description: Percentage of Participants achieving predefined antibody threshold levels for Pertussis Toxoid (PT) ≥5 ELISA units per milliliter (EU/mL), Filamentous Haemagglutinin (FHA) ≥5 or ≥7.82 EU/mL, and Pertactin (PRN) ≥5 EU/mL, ≥10.0 Milli-International Units Per Milliliter (mIU/mL) for Hepatitis B, Haemophilus Influenzae type b (Hib) 0.15 μg/ml, 0.01 or 0.1 IU/mL for Diphtheria, 0.1 IU/mL for Tetanus, and ≥1:8 titer for Polio (Type 1, 2, and 3) with the corresponding 95% CI for antigens are presented.
Time Frame: One month after the infant series (6 months of age) and after the toddler dose (12 months of age)
Population: Evaluable immunogenicity (per protocol) population who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate postinfant antibody concentration/titer for the given concomitant antigen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC After 2-Dose Infant Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 3 and 5 months of age (infant series).
- 7vPnC After 2-Dose Infant Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 3 and 5 months of age (infant series).
- 13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 11 months of age (toddler dose).
- 7vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 11 months of age (toddler dose).
Arm/Group | 13vPnC After 2-Dose Infant Series | 7vPnC After 2-Dose Infant Series | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 275 | 279 | 254 | 261
percentage of participants
  Pertussis, PT ≥5 EU/mL (n=250,272,235,219) | 99.6 [97.8 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.4 to 100.0] | 100.0 [98.3 to 100.0]
  Pertussis, FHA ≥5 EU/mL (n=243,272,229,214) | 100.0 [98.5 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.4 to 100.0] | 100.0 [98.3 to 100.0]
  Pertussis, FHA ≥7.82 EU/mL (n=243,272,229,214) | 100.0 [98.5 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.4 to 100.0] | 100.0 [98.3 to 100.0]
  Pertactin ≥5 EU/mL (n=248,270,234,217) | 100.0 [98.5 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.4 to 100.0] | 100.0 [98.3 to 100.0]
  Hepatitis B ≥ 10.0 mIU/mL | 93.8 [90.2 to 96.3] | 93.1 [89.5 to 95.8] | 98.40 [96.00 to 99.60] | 98.80 [96.60 to 99.80]
  Haemophilus Influenzae type b 0.15 μg/ml | 87.0 [82.0 to 91.1] | 90.3 [86.1 to 93.5] | 99.6 [97.7 to 100.0] | 98.2 [95.4 to 99.5]
  Haemophilus Influenzae type b 1.0 μg/ml | 49.9 [42.7 to 56.0] | 48.7 [42.6 to 54.9] | 96.2 [92.9 to 98.2] | 92.2 [87.8 to 95.4]
  Diptheria 0.01 IU/mL (n=207,240,164,190) | 100.0 [98.2 to 100.0] | 100.0 [98.5 to 100.0] | 100.0 [97.8 to 100.0] | 100.0 [98.1 to 100.0]
  Diptheria 0.1 IU/mL (n=207,240,164,190) | 92.8 [88.3 to 95.9] | 96.3 [93.0 to 98.3] | 100.0 [97.8 to 100] | 100.0 [98.1 to 100.0]
  Tetanus 0.1 IU/mL (n=155,214,125,96) | 94.2 [89.3 to 97.3] | 92.5 [88.1 to 95.7] | 97.6 [93.1 to 99.5] | 93.8 [86.9 to 97.7]
  Polio, Type 1 ≥1:8 | 99.5 [97.3 to 100.0] | 99.6 [97.9 to 100.0] | 100.0 [97.9 to 100.0] | 100.0 [98.0 to 100.0]
  Polio, Type 2 ≥1:8 | 95.6 [91.8 to 98.0] | 96.6 [93.6 to 98.4] | 100.0 [97.6 to 100.0] | 100.0 [97.9 to 100.0]
  Polio, Type 3 ≥1:8 | 99.5 [97.3 to 100.0] | 98.9 [96.7 to 99.8] | 100.0 [97.6 to 100.0] | 100.0 [97.9 to 100.0]
  Pertussis, PT (infant ≥16; Toddler ≥21) EU/mL | 95.2 [91.8 to 97.5] | 95.2 [92.0 to 97.4] | 92.8 [88.7 to 95.7] | 95.4 [91.8 to 97.8]
  Pertussis, FHA (Infant ≥31; Toddler ≥162) EU/mL | 94.7 [91.0 to 97.1] | 95.6 [92.4 to 97.7] | 95.2 [91.6 to 97.6] | 95.3 [91.6 to 97.7]
  Pertactin (Infant ≥40; Toddler ≥106) EU/mL | 91.9 [87.8 to 95.0] | 95.2 [91.9 to 97.4] | 94.9 [91.2 to 97.3] | 95.4 [91.7 to 97.8]
Statistical Analysis 1: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Pertussis PT the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥5 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lowest limit of the 2-sided 95% CI for the difference between the two groups was > -10%; Difference = -0.4, 95% CI [-2.2 to 1.0]
Statistical Analysis 2: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Pertussis PT the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥16 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-4.0 to 3.8]
Statistical Analysis 3: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Pertussis FHA the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥5 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-1.6 to 1.4]
Statistical Analysis 4: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Pertussis FHA the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥7.82 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-1.6 to 1.4]
Statistical Analysis 5: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Pertussis FHA the difference in percentages between the two groups ( 13vPnC - 7vPnC) at ≥31 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -0.90, 95% CI [-5.0 to 2.9]
Statistical Analysis 6: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Pertactin the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥5 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-1.5 to 1.4]
Statistical Analysis 7: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Pertactin the difference in percentages between the two groups ( 13vPnC - 7vPnC) at ≥40 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -3.2, 95% CI [-7.8 to 1.0]
Statistical Analysis 8: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For hepatitis B the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥10.0 mIU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.7, 95% CI [-3.6 to 5.0]
Statistical Analysis 9: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Haemophilus influenzae type b the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.15 μg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -3.2, 95% CI [-9.1 to 2.4]
Statistical Analysis 10: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Haemophilus influenzae type b the difference in percentages between the two groups (13vPnC - 7vPnC) at 1.0 μg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.7, 95% CI [-8.2 to 9.5]
Statistical Analysis 11: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Diptheria the difference in percentages between the two groups ( 13vPnC - 7vPnC) at 0.01 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-1.8 to 1.6]
Statistical Analysis 12: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Diptheria the difference in percentage between the two groups ( 13vPnC - 7vPnC) at 0.1 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -3.5, 95% CI [-8.3 to 0.8]
Statistical Analysis 13: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Tetanus the difference in percentage between the two groups ( 13vPnC - 7vPnC) at 0.1 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 1.7, 95% CI [-3.9 to 7.1]
Statistical Analysis 14: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Polio Type 1 the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥1:8 threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -0.1, 95% CI [-2.3 to 1.7]
Statistical Analysis 15: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Polio Type 2 the difference in percentage between the two groups ( 13vPnC - 7vPnC) at ≥1:8 threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -1.0, 95% CI [-5.0 to 2.8]
Statistical Analysis 16: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Polio Type 3 the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥1:8 threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.7, 95% CI [-1.6 to 2.9]
Statistical Analysis 17: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-1.6 to 1.7]
Statistical Analysis 18: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Pertussis PT the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥21 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -2.7, 95% CI [-7.3 to 1.8]
Statistical Analysis 19: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 3, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-1.6 to 1.7]
Statistical Analysis 20: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 3, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-1.6 to 1.7]
Statistical Analysis 21: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Pertussis FHA the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥162 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -0.1, 95% CI [-4.3 to 4.1]
Statistical Analysis 22: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 3, analysis 6]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-1.6 to 1.7]
Statistical Analysis 23: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Pertactin the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥106 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -0.5, 95% CI [-4.7 to 3.7]
Statistical Analysis 24: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 3, analysis 8]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = -0.4, 95% CI [-3.0 to 2.0]
Statistical Analysis 25: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Haemophilus influenzae type b the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.15 μg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 1.4, 95% CI [-0.8 to 4.2]
Statistical Analysis 26: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Haemophilus influenzae type b the difference in percentage between the two groups (13vPnC - 7vPnC) at 1.0 μg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 4.0, 95% CI [-0.4 to 8.7]
Statistical Analysis 27: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Diphtheria the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.01 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-2.3 to 2.0]
Statistical Analysis 28: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Diphtheria the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.1 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-2.3 to 2.0]
Statistical Analysis 29: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Tetanus the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.1 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 3.8, 95% CI [-1.7 to 10.9]
Statistical Analysis 30: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Polio Type 1 the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥1:8 threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-2.4 to 2.1]
Statistical Analysis 31: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Polio Type 2 the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥1:8 threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-2.4 to 2.1]
Statistical Analysis 32: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Polio Type 3 the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥1:8 threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference = 0.0, 95% CI [-2.4 to 2.1]

4. Primary Outcome: Geometric Mean Antibody Concentration (GMC) of Pertussis in the 13vPnC Group Relative to the 7vPnC Group After the 2-Dose Infant Series and After the Toddler Dose
Description: GMC of Pertussis (PT, FHA, PRN) were measured using an anti-Bordetella pertussis enzyme-linked immunosorbent assay (ELISA). Results were recorded in ELISA units per milliliter (EU/mL)
Time Frame: one month after infant series dose 2 (6 months of age) and after the toddler dose (12 months of age)
Population: Evaluable immunogenicity (per protocol) population adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Groups:
- 13vPnC After 2-Dose Infant Series: Subjects received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 3 and 5 months of age (infant series).
- 7vPnC After 2-Dose Infant Series: Subjects received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 3 and 5 months of age (infant series).
- 13vPnC After Toddler Dose: Subjects received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 11 months of age (toddler dose).
- 7vPnC After Toddler Dose: Subjects received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 11 months of age (toddler dose).
Arm/Group | 13vPnC After 2-Dose Infant Series | 7vPnC After 2-Dose Infant Series | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 275 | 279 | 254 | 261
EU/mL
  Pertussis FHA | 102.87 [94.35 to 112.16] | 105.17 [97.25 to 113.73] | 463.23 [425.19 to 504.67] | 456.55 [415.06 to 502.18]
  Pertussis PT | 50.01 [45.82 to 54.58] | 48.44 [44.71 to 52.49] | 60.89 [55.61 to 66.67] | 64.53 [59.13 to 70.42]
  Pertussis PRN | 167.76 [149.54 to 188.18] | 166.19 [150.28 to 183.78] | 339.30 [309.16 to 372.38] | 361.70 [328.59 to 398.14]
Statistical Analysis 1: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Pertussis FHA the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lower bound of the 2-sided, 95% CI for the GMC/GMT ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 0.98, 95% CI [0.87 to 1.10]
Statistical Analysis 2: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Pertussis PT the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 1.03, 95% CI [0.92 to 1.16]
Statistical Analysis 3: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Pertussis PRN the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 1.01, 95% CI [0.87 to 1.17]
Statistical Analysis 4: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Pertussis FHA the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 1.01, 95% CI [0.89 to 1.15]
Statistical Analysis 5: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Pertussis PT the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.94, 95% CI [0.83 to 1.07]
Statistical Analysis 6: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Pertussis PRN the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.94, 95% CI [0.82 to 1.07]

5. Other Pre Specified Outcome: Percentage of Subjects Achieving Antibody Titer (OPA) ≥1:8 in 13vPnC Group After the 2-Dose Infant Series and the Toddler Dose
Description: Percentage of subjects achieving functional antibody titer ≥1:8 as measured by opsonophagocytic activity assay (OPA) along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. (This is not a geometric mean comparison as suggested by the table row heading).
Time Frame: one month after infant series dose 2 and after the toddler dose
Population: OPAs were done in a subset of approximately 100 subjects (range 90-100 per serotype) in the 13vPnC group
Measure: Geometric Mean (95% Confidence Interval); unit: % Achieving OPA Titer ≥1:8
Arm/Group | 13vPnC After 2-Dose Infant Series | 13vPnC After Toddler Dose
Number analyzed (Participants) | 100 | 100
% Achieving OPA Titer ≥1:8
  Common Serotypes - Serotype 4 | 100.0 [96.3 to 100.0] | 100.0 [95.8 to 100.0]
  Common Serotypes - Serotype 6B | 90.0 [82.4 to 95.1] | 99.0 [94.3 to 100.0]
  Common Serotypes - Serotype 9V | 100.0 [96.3 to 100.0] | 100.0 [96.1 to 100.0]
  Common Serotypes - Serotype 14 | 100.0 [96.3 to 100.0] | 100.0 [96.2 to 100.0]
  Common Serotypes - Serotype 18C | 97.0 [91.4 to 99.4] | 100.0 [96.3 to 100.0]
  Common Serotypes - Serotype 19F | 96.0 [90.1 to 98.9] | 97.9 [92.7 to 99.7]
  Common Serotypes - Serotype 23F | 97.0 [91.4 to 99.4] | 100.0 [96.3 to 100.0]
  Additional Serotypes - Serotype 1 | 94.8 [88.3 to 98.3] | 100.0 [96.2 to 100.0]
  Additional Serotypes - Serotype 3 | 99.0 [94.6 to 100.0] | 100.0 [96.2 to 100.0]
  Additional Serotypes - Serotype 5 | 96.0 [90.0 to 98.9] | 100.0 [96.1 to 100.0]
  Additional Serotypes - Serotype 6A | 95.9 [89.9 to 98.9] | 100.0 [96.2 to 100.0]
  Additional Serotypes - Serotype 7F | 100.0 [96.4 to 100.0] | 100.0 [96.2 to 100.0]
  Additional Serotypes - Serotype 19A | 95.6 [89.0 to 98.8] | 100.0 [96.0 to 100.0]

6. Other Pre Specified Outcome: Geometric Mean Antibody Titer (OPA) in 13vPnC Group After the 2-Dose Infant Series and the Toddler Dose
Description: Antibody functionality/geometric mean titer (GMT) as measured by opsonophagocytic activity assay(OPA) for7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: one month after infant series dose 2 and after the toddler dose
Population: OPAS were done in a subset of approximately 100 subjects (range 90-100 per serotype) in the 13vPnC group
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 13vPnC After 2-Dose Infant Series | 13vPnC After Toddler Dose
Number analyzed (Participants) | 100 | 100
Titers
  Common Serotypes - Serotype 4 | 526.69 [431.88 to 642.32] | 1276.21 [1025.09 to 1588.85]
  Common Serotypes - Serotype 6B | 191.34 [133.35 to 274.55] | 2383.31 [1850.47 to 3069.57]
  Common Serotypes - Serotype 9V | 3585.80 [2787.34 to 4612.99] | 16384.00 [13066.97 to 20543.06]
  Common Serotypes - Serotype 14 | 1882.96 [1446.51 to 2451.10] | 1903.89 [1580.90 to 2292.88]
  Common Serotypes - Serotype 18C | 294.48 [221.80 to 390.98] | 1324.41 [1063.57 to 1649.22]
  Common Serotypes - Serotype 19F | 222.86 [170.46 to 291.37] | 391.97 [296.34 to 518.46]
  Common Serotypes - Serotype 23F | 487.51 [356.25 to 667.13] | 3679.67 [2971.61 to 4556.44]
  Additional Serotypes - Serotype 1 | 62.63 [47.59 to 82.41] | 294.07 [226.88 to 381.15]
  Additional Serotypes - Serotype 3 | 176.07 [144.89 to 213.96] | 504.66 [435.71 to 584.53]
  Additional Serotypes - Serotype 5 | 127.11 [99.36 to 162.60] | 333.24 [274.24 to 404.94]
  Additional Serotypes - Serotype 6A | 541.81 [392.09 to 748.68] | 2217.29 [1821.95 to 2698.42]
  Additional Serotypes - Serotype 7F | 5914.33 [4710.83 to 7425.30] | 14886.35 [12560.25 to 17643.22]
  Additional Serotypes - Serotype 19F | 157.59 [118.91 to 208.84] | 1415.08 [1140.56 to 1755.66]

7. Primary Outcome: Geometric Mean Antibody Concentration (GMC) for Hepatitis B in the 13vPnC Group Relative to the 7vPnC Group After the 2-Dose Infant Series and After Toddler Dose
Description: GMC of anti-hepatitis B surface antigen (HBsAg)using an Food and Drug Administration (FDA) approved in vitro diagnostic kit.
Time Frame: One month after the infant series (6 months of age) and the toddler dose (12 months of age)
Population: Evaluable immunogenicity (per protocol) population had valid and determinate assay results, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: mIU/mL
Groups:
- 13vPnC After Toddler Dose: Participants received one single 0.5 mL 13vPnC coadministered with Infanrix hexa at 11 months of age (toddler dose).
- 7vPnC After Toddler Dose: Participants received one single 0.5 mL 7vPnC coadministered with Infanrix hexa at 11 months of age (toddler dose).
Arm/Group | 13vPnC After 2-Dose Infant Series | 7vPnC After 2-Dose Infant Series | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 273 | 276 | 252 | 255
mIU/mL | 260.46 [214.47 to 316.31] | 272.67 [220.83 to 336.68] | 1655.30 [1343.30 to 2039.77] | 2284.95 [1878.82 to 2778.88]
Statistical Analysis 1: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Hepatitis b the geometric mean concentration (GMC) ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lower bound of the 2-sided, 95% CI for the geometric mean concentration (GMC)/geometric mean titer (GMT) ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 0.96, 95% CI [0.72 to 1.27]
Statistical Analysis 2: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Hepatitis b the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.72, 95% CI [0.54 to 0.96]

8. Primary Outcome: Geometric Mean Antibody Concentration (GMC) of Haemophilus Influenzae Type b (Hib) in the 13vPnC Group Relative to the 7vPnC Group After the 2-Dose Infant Series and After the Toddler Dose
Description: GMC for Hib polyribosylribitol phosphate as measured by ELISA, expressed in micrograms per milliliter (μg/mL).
Time Frame: one month after infant series dose 2 (6 months of age) and after the toddler dose (12 months of age)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC After 2-Dose Infant Series | 7vPnC After 2-Dose Infant Series | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 231 | 267 | 235 | 218
μg/mL | 0.99 [0.80 to 1.21] | 1.00 [0.83 to 1.20] | 9.09 [7.80 to 10.60] | 8.85 [7.37 to 10.62]
Statistical Analysis 1: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; or Haemophilus influenzae type b the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.99, 95% CI [0.75 to 1.30]
Statistical Analysis 2: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Haemophilus influenzae type b the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 1.03, 95% CI [0.81 to 1.30]

9. Primary Outcome: Geometric Mean Antibody Concentration (GMC) of Diptheria and Tetanus in the 13vPnC Group Relative to the 7vPnC Group After the 2-Dose Infant Series and After the Toddler Dose
Description: GMC of anti-diphtheria and anti-tetanus toxoids as measured by ELISA (IU/mL).
Time Frame: one month after infant series dose 2 (6 months of age) and after the toddler dose (12 months of age)
Population: Evaluable immunogenicity (per protocol) population had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate antibody concentration/titer for the specified concomitant antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 13vPnC After 2-Dose Infant Series | 7vPnC After 2-Dose Infant Series | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 275 | 279 | 254 | 261
IU/mL
  Diptheria (n=207,240,164,190) | 0.52 [0.46 to 0.60] | 0.67 [0.59 to 0.76] | 2.77 [2.45 to 3.13] | 3.71 [3.28 to 4.20]
  Tetanus (n=155,214,125,96) | 0.53 [0.45 to 0.63] | 0.63 [0.53 to 0.74] | 2.62 [2.12 to 3.25] | 2.09 [1.56 to 2.81]
Statistical Analysis 1: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For diphtheria toxoid the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.78, 95% CI [0.65 to 0.94]
Statistical Analysis 2: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Tetanus the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.85, 95% CI [0.67 to 1.08]
Statistical Analysis 3: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For diphtheria toxoid the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.75, 95% CI [0.63 to 0.89]
Statistical Analysis 4: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Tetanus the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 1.25, 95% CI [0.88 to 1.79]

10. Primary Outcome: Geometric Mean Antibody Concentration (GMC) of Polio Types 1, 2, and 3 in the 13vPnC Group Relative to the 7vPnC Group After the 2-Dose Infant Series and After the Toddler Dose
Description: GMC of Polio as measured using a polio in vitro plaque neutralization.
Time Frame: one month after infant series dose 2 (6 months of age) and after the toddler dose (12 months of age)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 13vPnC After 2-Dose Infant Series | 7vPnC After 2-Dose Infant Series | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 275 | 279 | 254 | 261
Titers
  Polio Type 1 (n=207,262,156,179) | 180.72 [154.31 to 211.64] | 207.17 [178.64 to 240.25] | 924.52 [782.71 to 1092.03] | 1348.04 [1163.56 to 1561.77]
  Polio Type 2 (n=205,262,153,175) | 123.74 [102.68 to 149.13] | 130.39 [109.96 to 154.63] | 1141.62 [958.68 to 1359.47] | 1340.51 [1147.88 to 1565.48]
  Polio Type 3 (n=205,262,153,178) | 397.32 [327.00 to 482.76] | 452.14 [382.57 to 534.35] | 1567.64 [1289.72 to 1905.45] | 2421.31 [2072.82 to 2828.39]
Statistical Analysis 1: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Polio Type 1 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.87, 95% CI [0.70 to 1.08]
Statistical Analysis 2: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Polio Type 2 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.95, 95% CI [0.74 to 1.22]
Statistical Analysis 3: Comparison: 13vPnC After 2-Dose Infant Series vs 7vPnC After 2-Dose Infant Series; For Polio Type 3 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.88, 95% CI [0.68 to 1.13]
Statistical Analysis 4: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Polio Type 1 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.69, 95% CI [0.55 to 0.86]
Statistical Analysis 5: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Polio Type 2 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.85, 95% CI [0.68 to 1.07]
Statistical Analysis 6: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Polio Type 3 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.65, 95% CI [0.51 to 0.83]

11. Primary Outcome: Percentage of Participants Achieving an Antibody Level of ≥0.35 μg/mL in the 13vPnC Group After the 2-Dose Infant Series and Before the Toddler Dose
Description: Percentages of Participants achieving World Health Organization (WHO) predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: one month after infant series dose 2 (6 months of age) and before the toddler dose (11 months of age)
Population: The evaluable pneumococcal immunogenicity (per protocol) population was the primary analysis population consisting of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC Before Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 11 months of age (toddler dose).
Arm/Group | 13vPnC After 2-Dose Infant Series | 13vPnC Before Toddler Dose
Number analyzed (Participants) | 265 | 265
percentage of participants
  Common Serotypes - Serotype 4 | 96.6 [93.6 to 98.4] | 66.9 [60.6 to 72.9]
  Common Serotypes - Serotype 6B | 58.4 [52.2 to 64.4] | 76.3 [70.3 to 81.6]
  Common Serotypes - Serotype 9V | 94.7 [91.2 to 97.1] | 70.5 [64.2 to 76.2]
  Common Serotypes - Serotype 14 | 94.2 [90.6 to 96.7] | 94.4 [90.6 to 97.0]
  Common Serotypes - Serotype 18C | 92.4 [88.5 to 95.3] | 53.0 [46.4 to 59.5]
  Common Serotypes - Serotype 19F | 95.1 [91.7 to 97.3] | 92.4 [88.2 to 95.4]
  Common Serotypes - Serotype 23F | 68.6 [62.6 to 74.1] | 32.3 [26.4 to 38.7]
  Additional Serotypes - Serotype 1 | 96.6 [93.6 to 98.4] | 83.4 [78.0 to 87.9]
  Additional Serotypes - Serotype 3 | 92.8 [89.0 to 95.6] | 30.8 [24.9 to 37.1]
  Additional Serotypes - Serotype 5 | 91.6 [87.5 to 94.6] | 87.3 [82.4 to 91.3]
  Additional Serotypes - Serotype 6A | 86.5 [81.8 to 90.4] | 86.4 [81.4 to 90.5]
  Additional Serotypes - Serotype 7F | 98.5 [96.2 to 99.6] | 90.7 [86.3 to 94.1]
  Additional Serotypes - Serotype 19A | 98.5 [96.1 to 99.6] | 96.2 [92.9 to 98.2]

12. Primary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody in 13vPnC Group After the 2-Dose Infant Series and Before Toddler Dose
Description: Antibody GMC for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after infant series dose 2 (6 months of age) and before the toddler dose (11 months of age)
Population: Evaluable pneumococcal immunogenicity (per protocol) had valid and determinate assay results, and had no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC After 2-Dose Infant Series | 13vPnC Before Toddler Dose
Number analyzed (Participants) | 265 | 265
μg/mL
  Common Serotypes - Serotype 4 | 2.38 [2.11 to 2.67] | 0.53 [0.48 to 0.59]
  Common Serotypes - Serotype 6B | 0.41 [0.36 to 0.47] | 0.61 [0.54 to 0.69]
  Common Serotypes - Serotype 9V | 1.68 [1.51 to 1.86] | 0.48 [0.43 to 0.52]
  Common Serotypes - Serotype 14 | 2.84 [2.44 to 3.31] | 2.03 [1.79 to 2.30]
  Common Serotypes - Serotype 18C | 1.72 [1.54 to 1.93] | 0.35 [0.32 to 0.39]
  Common Serotypes - Serotype 19F | 3.42 [2.95 to 3.97] | 0.94 [0.83 to 1.06]
  Common Serotypes - Serotype 23F | 0.61 [0.53 to 0.71] | 0.26 [0.23 to 0.29]
  Additional Serotypes - Serotype 1 | 2.30 [2.03 to 2.60] | 0.68 [0.61 to 0.75]
  Additional Serotypes - Serotype 3 | 1.15 [1.04 to 1.28] | 0.25 [0.22 to 0.27]
  Additional Serotypes - Serotype 5 | 1.27 [1.14 to 1.41] | 0.88 [0.80 to 0.97]
  Additional Serotypes - Serotype 6A | 1.17 [1.02 to 1.33] | 0.81 [0.72 to 0.92]
  Additional Serotypes - Serotype 7F | 2.06 [1.88 to 2.26] | 0.76 [0.70 to 0.82]
  Additional Serotypes - Serotype 19F | 2.87 [2.55 to 3.24] | 1.20 [1.06 to 1.35]

13. Secondary Outcome: Percentage of Participants Achieving an Antibody Level of ≥0.35 μg/mL in the 13vPnC Relative to the 7vPnC Group After the Toddler Dose
Description: Percentages of Participants achieving WHO predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after the toddler dose (12 months of age)
Population: Evaluable pneumococcal immunogenicity (per protocol) population had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate IgG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 246 | 249
percentage of participants
  Common Serotypes - Serotype 4 (n=244,245) | 100.0 [98.5 to 100.0] | 100.0 [98.5 to 100.0]
  Common Serotypes - Serotype 6B (n=243,243) | 100.0 [98.5 to 100.0] | 100.0 [98.5 to 100.0]
  Common Serotypes - Serotype 9V (n=235,248) | 100.0 [98.4 to 100.0] | 100.0 [98.5 to 100.0]
  Common Serotypes - Serotype 14 (n=237,240) | 99.6 [97.7 to 100.0] | 99.6 [97.7 to 100.0]
  Common Serotypes - Serotype 18C (n=245,245) | 99.2 [97.1 to 99.9] | 99.6 [97.8 to 100.0]
  Common Serotypes - Serotype 19F (n=243,245) | 98.8 [96.4 to 99.7] | 98.4 [95.9 to 99.6]
  Common Serotypes - Serotype 23F (n=240,243) | 99.2 [97.0 to 99.9] | 98.8 [96.4 to 99.7]
  Additional Serotypes - Serotype 1 (n=244,240) | 99.6 [97.7 to 100.0] | 3.3 [1.4 to 6.5]
  Additional Serotypes - Serotype 3 (n=245,218) | 93.9 [90.1 to 96.5] | 6.7 [3.9 to 10.6]
  Additional Serotypes - Serotype 5 (n=245,243) | 100.0 [98.5 to 100.0] | 70.2 [63.6 to 76.2]
  Additional Serotypes - Serotype 6A (n=243,243) | 99.6 [97.7 to 100.0] | 86.4 [81.5 to 90.5]
  Additional Serotypes - Serotype 7F (n=242,243) | 99.6 [97.7 to 100.0] | 4.9 [2.6 to 8.5]
  Additional Serotypes - Serotype 19A (n=241,241) | 100.0 [98.5 to 100.0] | 99.6 [97.7 to 100.0]

14. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody in 13vPnC Relative to 7vPnC Group After the Toddler Dose
Description: as for outcome 12
Time Frame: One month after toddler dose (12 months of age)
Population: Evaluable pneumococcal immunogenicity (per protocol) had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate antibody concentration for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- 13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 12 months of age (toddler dose).
- 7vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 12 months of age (toddler dose).
Arm/Group | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 246 | 249
μg/mL
  Common Serotypes - Serotype 4 (n=244,245) | 4.77 [4.29 to 5.30] | 7.08 [6.41 to 7.83]
  Common Serotypes - Serotype 6B (n=243,243) | 10.00 [8.79 to 11.38] | 10.39 [9.14 to 11.82]
  Common Serotypes - Serotype 9V (n=235,248) | 3.02 [2.74 to 3.32] | 4.10 [3.72 to 4.51]
  Common Serotypes - Serotype 14 (n=237,240) | 10.30 [9.26 to 11.47] | 11.99 [10.77 to 13.35]
  Common Serotypes - Serotype 18C (n=245,247) | 2.83 [2.55 to 3.14] | 4.26 [3.85 to 4.70]
  Common Serotypes - Serotype 19F (n=243,245) | 9.01 [7.84 to 10.36] | 8.06 [7.06 to 9.21]
  Common Serotypes - Serotype 23F (n=244,245) | 3.43 [3.02 to 3.88] | 4.87 [4.30 to 5.51]
  Additional Serotypes - Serotype 1 (n=244,240) | 5.76 [5.12 to 6.47] | 0.03 [0.03 to 0.04]
  Additional Serotypes - Serotype 3 (n=245,240) | 1.22 [1.09 to 1.35] | 0.07 [0.06 to 0.08]
  Additional Serotypes - Serotype 5 (n=245,218) | 3.59 [3.25 to 3.96] | 0.56 [0.49 to 0.64]
  Additional Serotypes - Serotype 6A (n=243,243) | 6.78 [6.04 to 7.61] | 1.42 [1.21 to 1.66]
  Additional Serotypes - Serotype 7F (n=242,243) | 4.31 [3.94 to 4.72] | 0.04 [0.04 to 0.05]
  Additional Serotypes - Serotype 19F (n=241,241) | 9.81 [8.82 to 10.92] | 4.24 [3.85 to 4.67]

ADVERSE EVENTS:
Groups:
- 13vPnC Infant Series: Participants received one single 0.5mL dose of 13vPnC coadministered with Infanrix hexa at 3 and 5 months. Adverse events were collected from dose 1 to approximately one month after dose 2.
- 7vPnC Infant Series: Participants received one single 0.5mL dose of 7vPnC coadministered with Infanrix hexa at 3 and 5 months. Adverse events were collected from dose 1 to approximately one month after dose 2.
- 13vPnC Post-Infant Series: Participants received one single 0.5mL dose of 13vPnC coadministered with Infanrix hexa at 3 and 5 months. Adverse events were collected from approximately one month after dose 2 to toddler dose.
- 7vPnC Post-Infant Series: Participants received one single 0.5mL dose of 7vPnC coadministered with Infanrix hexa at 3 and 5 months. Adverse events were collected from approximately one month after dose 2 to toddler dose.
- 13vPnC Toddler Series: Participants received one single 0.5mL dose of 13vPnC at 11 months of age. Adverse events were collected for approximately one month after toddler dose.
- 7vPnC Toddler Series: Participants received one single 0.5mL dose of 7vPnC at 11 months of age. Adverse events were collected for approximately one month after toddler dose.
- 13vPnC 6-Month Follow-up: Participants received one single 0.5mL dose of 13vPnC coadministered with Infanrix hexa at 3 and 5 months (infant series) and 11 months of age (toddler dose). Adverse events were collected for approximately six months after last visit.
- 7vPnC 6-Month Follow-up: Participants received one single 0.5mL dose of 7vPnC coadministered with Infanrix hexa at 3 and 5 months (infant series) and 11 months of age (toddler dose). Adverse events were collected for approximately six months after last visit.
Arm/Group | 13vPnC Infant Series | 7vPnC Infant Series | 13vPnC Post-Infant Series | 7vPnC Post-Infant Series | 13vPnC Toddler Series | 7vPnC Toddler Series | 13vPnC 6-Month Follow-up | 7vPnC 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 6/303 | 10/303 | 8/294 | 11/291 | 3/287 | 1/282 | 9/290 | 11/288
Other Adverse Events (participants affected / at risk) | 188/303 | 183/303 | 96/294 | 90/291 | 165/287 | 170/282 | 1/290 | 0/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Infant Series (N=303) | 7vPnC Infant Series (N=303) | 13vPnC Post-Infant Series (N=294) | 7vPnC Post-Infant Series (N=291) | 13vPnC Toddler Series (N=287) | 7vPnC Toddler Series (N=282) | 13vPnC 6-Month Follow-up (N=290) | 7vPnC 6-Month Follow-up (N=288)
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis orbital (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Crying (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased activity (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 4
Gastroenteritis adenovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokinesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infantile spasms (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Kawasaki's disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningism (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otits media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelizaeus-Merzbacher disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Infant Series (N=303) | 7vPnC Infant Series (N=303) | 13vPnC Post-Infant Series (N=294) | 7vPnC Post-Infant Series (N=291) | 13vPnC Toddler Series (N=287) | 7vPnC Toddler Series (N=282) | 13vPnC 6-Month Follow-up (N=290) | 7vPnC 6-Month Follow-up (N=288)
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 75/234 | 73/243 | 0/0 | 0/0 | 94/199 | 83/188 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 65/214 | 79/215 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 6/224 | 8/231 | 0/0 | 0/0 | 14/164 | 9/153 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 9/199 | 10/199 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Induration (Any) (Skin and subcutaneous tissue disorders) | 44/232 | 47/240 | 0/0 | 0/0 | 50/175 | 45/165 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Induration (Any) (Skin and subcutaneous tissue disorders) | 51/207 | 60/209 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Induration (Mild) (Skin and subcutaneous tissue disorders) | 41/232 | 44/240 | 0/0 | 0/0 | 46/174 | 35/161 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Induration (Mild) (Skin and subcutaneous tissue disorders) | 45/207 | 55/208 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 8/223 | 7/229 | 0/0 | 0/0 | 12/160 | 16/157 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 11/198 | 10/195 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/222 | 0/229 | 0/0 | 0/0 | 0/159 | 0/152 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/197 | 0/194 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Erythema (Any) (Skin and subcutaneous tissue disorders) | 60/233 | 65/245 | 0/0 | 0/0 | 65/178 | 63/174 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Erythema (Any) (Skin and subcutaneous tissue disorders) | 67/213 | 73/212 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 56/233 | 60/244 | 0/0 | 0/0 | 58/178 | 53/172 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 60/211 | 68/211 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 6/222 | 7/231 | 0/0 | 0/0 | 12/160 | 17/156 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 11/200 | 7/195 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/222 | 0/229 | 0/0 | 0/0 | 0/159 | 0/152 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/197 | 0/194 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Fever ≥38°C but ≤39°C (General disorders) | 103/247 | 95/246 | 0/0 | 0/0 | 130/204 | 103/197 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Fever ≥38°C but ≤39°C (General disorders) | 126/227 | 137/226 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Fever >39°C but ≤40°C (General disorders) | 8/224 | 11/233 | 0/0 | 0/0 | 16/167 | 20/160 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Fever >39°C but ≤40°C (General disorders) | 14/204 | 14/201 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Fever >40°C (General disorders) | 0/222 | 0/230 | 0/0 | 0/0 | 0/160 | 1/152 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Fever >40°C (General disorders) | 0/198 | 0/195 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Decreased appetite (General disorders) | 87/246 | 85/248 | 0/0 | 0/0 | 103/198 | 113/197 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Decreased appetite (General disorders) | 104/220 | 99/218 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Irritability (General disorders) | 188/258 | 165/259 | 0/0 | 0/0 | 165/221 | 170/227 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Irritability (General disorders) | 185/245 | 183/243 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Increased sleep (General disorders) | 177/269 | 178/276 | 0/0 | 0/0 | 105/195 | 107/196 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Increased sleep (General disorders) | 129/226 | 131/232 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Decreased sleep (General disorders) | 96/244 | 88/242 | 0/0 | 0/0 | 64/180 | 61/171 | 0/0 | 0/0 — Dose 1 Infant Series & Toddler Dose
Decreased sleep (General disorders) | 89/222 | 89/213 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 5 | 1 | 0 | 0 | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid cyst (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 4 | 1 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 12 | 2 | 5/5 | 8 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 5 | 1 | 3 | 4 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perianal erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 24 | 23 | 33 | 34 | 25 | 16 | 0 | 0
Irritability (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 13 | 10 | 8 | 12 | 4 | 7 | 0 | 0
Rhinitis (Infections and infestations) | 11 | 10 | 6 | 4 | 9 | 5 | 0 | 0
Bronchiolitis (Infections and infestations) | 8 | 9 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 8 | 6 | 16 | 7 | 2 | 11 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 5 | 4 | 8 | 3 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 6 | 0 | 3 | 1 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 4 | 4 | 5 | 5 | 1 | 0 | 0
Exanthema subitum (Infections and infestations) | 4 | 3 | 16 | 22 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 4 | 2 | 7 | 7 | 6 | 7 | 0 | 0
Influenza (Infections and infestations) | 1 | 5 | 1 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 3 | 8 | 5 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 3 | 5 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0
Viral skin infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Roseola (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 18 | 8 | 7 | 8 | 7 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 1 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 5 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1/1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.